CLINICAL TRIAL: NCT06029543
Title: Permian Health Women's Lung Health Study
Acronym: WLHS
Status: Not yet recruiting | Type: Observational
Sponsor: Permian Health Lung Institute (Other)
Collaborators: The Gambia Committee on Traditional Practices Affecting the Health of Women and Children (GAMCOTRAP) (Unknown)
Responsible Party: Sponsor
Other Study IDs: WLHS2023001
Record Dates: First submitted 2023-08-26; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: COPD; Lung Function Decreased; Alpha 1-Antitrypsin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; alpha 1-Antitrypsin Deficiency

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gambian Women: Gambian women aged 15 and older with lung function impairment as measured by spirometry

SUMMARY:
The goal of this cross-sectional observational study is to estimate the prevalence of lung function impairment as measured by spirometry in a population of Gambian women aged 15 and older. The main question[s] it aims to answer are:

* What is the prevalence of lung function impairment in Gambian women
* What is the prevalence of eosinophilic inflammation in Gambian women

Consenting participants will undergo

* Spirometry
* Fractional exhaled nitric oxide (FENO) testing
* α1-antitrypsin testing in patients with lung function impairment as assessed by spirometry

ELIGIBILITY:
Inclusion criteria:

* Self-identified female sex
* Age > 15 years: This age cutoff was chosen (as opposed to 18) because of the unique cultural norms and practices in the country where experiences and exposures occur at an earlier age than women in Western countries.

Exclusion criteria:

* Age < 15 years
* Non-resident household member
* Any acutely unwell individual
* Pregnancy
* Any known history of active pulmonary disease (including TB) on treatment.
* Individuals unable or unwilling to give consent.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Self-identified female sex
Study Population: All women older than 15 years in The Gambia
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of lung function Impairment as measured by spirometry | Through study completion, an average of 1 year
  Certified technicians will perform Spirometry testing to measure lung function parameters such as FEV1, FVC, and FEV1/FVC ratio. Results will be interpreted by two Pulmonologists using GLI reference equations and z-scores. Bronchodilator reversibility is defined as an improvement of over 10% in FEV1 after albuterol sulfate administration. Lung function impairment will be assessed based on z-scores, with normal lung function being z-scores greater than -1.645, mild impairment between -1.65 and -2.5, moderate impairment between -2.51 and -4, and severe impairment below -4.1.

SECONDARY OUTCOMES:
Prevalence of Type II (Eosinophilic) inflammation in Gambian Women | Through study completion, an average of 1 year
  FENO measurements will be taken using handheld devices called NIOX VERO. These devices are compliant with guidelines set by the American Thoracic Society and European Respiratory Society. To measure FENO, participants will be instructed to exhale into the device through a filtered mouthpiece. The exhaling process will be regulated to maintain a controlled flow rate and pressure for a duration of 10 seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Gamcotrap, Kanifing, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ale BM, Ozoh OB, Gadanya MA, Li Y, Harhay MO, Adebiyi AO, Adeloye D. Estimating the prevalence of COPD in an African country: evidence from southern Nigeria. J Glob Health Rep. 2022;6:e2022049. doi: 10.29392/001c.38200. Epub 2022 Sep 15. PMID 36185970
- [Background] Chan-Yeung M, Ait-Khaled N, White N, Ip MS, Tan WC. The burden and impact of COPD in Asia and Africa. Int J Tuberc Lung Dis. 2004 Jan;8(1):2-14. PMID 14974740
- [Background] Halbert RJ, Natoli JL, Gano A, Badamgarav E, Buist AS, Mannino DM. Global burden of COPD: systematic review and meta-analysis. Eur Respir J. 2006 Sep;28(3):523-32. doi: 10.1183/09031936.06.00124605. Epub 2006 Apr 12. PMID 16611654
- [Background] Stoller JK, Sandhaus RA, Turino G, Dickson R, Rodgers K, Strange C. Delay in diagnosis of alpha1-antitrypsin deficiency: a continuing problem. Chest. 2005 Oct;128(4):1989-94. doi: 10.1378/chest.128.4.1989. PMID 16236846
- [Background] Chapman KR, Chorostowska-Wynimko J, Koczulla AR, Ferrarotti I, McElvaney NG. Alpha 1 antitrypsin to treat lung disease in alpha 1 antitrypsin deficiency: recent developments and clinical implications. Int J Chron Obstruct Pulmon Dis. 2018 Jan 31;13:419-432. doi: 10.2147/COPD.S149429. eCollection 2018. PMID 29430176
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society statement: standards for the diagnosis and management of individuals with alpha-1 antitrypsin deficiency. Am J Respir Crit Care Med. 2003 Oct 1;168(7):818-900. doi: 10.1164/rccm.168.7.818. No abstract available. PMID 14522813